CLINICAL TRIAL: NCT01883414
Title: Feasibility Study: Evaluation of the Ulthera® System for Improvement of Surgical Scars.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources to manage trial; lack of efficacy.
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-136 Avram
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2014-03

CONDITIONS: Surgical Scar
Keywords: Ulthera, Ultherapy, Surgical scar, scar,
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Subjects randomized to Group A will receive Ultherapy™ treatment on the superior or lateral half of the scar.
  Interventions: Device: Ultherapy™
- Group B (Active Comparator): Subjects randomized to Group B will receive Ultherapy™ treatment on the inferior or medial half of the scar.
  Interventions: Device: Ultherapy™

INTERVENTIONS:
Device: Ultherapy™ — All subjects will receive an Ultherapy™ treatment at triple depth using the 4-4.5mm, 7- 3.0mm, 10-1.5mm transducers on one half of the scar and no treatment on the other half of the scar. Treatments will be provided to the defined scar area, treating with a density of lines that is equivalent to 30 lines per transducer per 2.5cm in scar length for a total of 90 lines in a 2.5cm X 2.5cm square area.

SUMMARY:
Up to 25 subjects will be enrolled. Enrolled subjects will received on Ulthera® treatment on one half of their surgical scar. Follow up visits will occur at 30, 90 and 180 days after treatment. Study images will be obtained before treatment, immediately after treatment and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, single-center, pilot clinical trial to evaluate the efficacy of the Ulthera® system to improve the appearance of scar tissue on the neck, abdomen or back. Changes from baseline of the Patient Observer Scar Assessment Scale score will be assessed at study follow-up visits. Images will be obtained prior to treatment and at each follow up visit. Patient satisfaction questionnaires will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 70 years.
2. Subject in good health.
3. Subjects will have regularly shaped surgical scars on the chest, abdomen or back that are at least 4 cm long, are no wider than 1 cm, and are at least 6 months old.
4. Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
5. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
6. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

   * Postmenopausal for at least 12 months prior to study;
   * Without a uterus and/or both ovaries; or
   * Bilateral tubal ligation at least six months prior to study enrollment.

Exclusion Criteria:

1. Presence of an active systemic or local skin disease that may affect wound healing.
2. Allergy to any pain medications used in the study (lidocaine, NSAIDs, narcotics, etc.)
3. Severe solar elastosis.
4. Open wounds or lesions in the area(s) to be treated.
5. Severe or cystic acne on the area(s) to be treated.
6. Presence of a metal stent or implant in the area(s) to be treated.
7. Inability to understand the protocol or to give informed consent.
8. Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within three months prior to study participation or during the study.
9. Intralesional kenalog in the past 6 months.
10. History of chronic drug or alcohol abuse.
11. History of autoimmune disease.
12. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
13. Subjects who anticipate the need for surgery or overnight hospitalization during the study.
14. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
15. Concurrent enrollment in any study involving the use of investigational devices or drugs.
16. Current smoker or history of smoking in the last year.
17. History of the following treatments in the area(s) to be treated:

    1. Skin tightening procedure within the past year;
    2. Injectable filler of any type within the past:

    i. 12 months for Hyaluronic acid fillers (e.g. Restylane) ii. 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse) iii. 24 months for Poly-L-Lactic acid fillers (e.g. Sculptra) iv. Ever for permanent fillers (e.g. Silicone, ArteFill) c. Neurotoxins within the past three months; d. Ablative resurfacing laser treatment; e. Nonablative, rejuvenative laser or light treatment within the past six months; f. Surgical dermabrasion or deep peels; g. Any history of contour threads.
18. History of using the following prescription medications:

    1. Accutane or other systemic retinoids within the past six months;
    2. Topical Retinoids within the past two weeks;
    3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix, etc.);
    4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.
    5. Subjects that are immunocompromised or are on immunosuppressive therapy
19. Subjects that are immunocompromised or are on immunosuppressive therapy
20. History of keloids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is improvement in appearance of scar tissue as determined by a masked, qualitative assessment of photographs at 90-days post-treatment time points comparing the treated to untreated side of the scar. | 90 days
  Masked assessors will compare baseline images to images obtained at the 90 day follow up time point in a blinded fashion.

SECONDARY OUTCOMES:
1. Improvement in POSAS score of the treated half of the scar as assessed by the observer using the Patient and Observer Scar Assessment Scale (POSAS) at 90-days post-treatment compared to baseline. | 90 Days
  The observer will complete the Patient and Observer Scar Assessment Scale (6 questions) prior to treatment and at each follow up visit on both halves of the scar (treated and untreated). Scores will be tabulated and compared for improvement at 90 days after treatment.
2. Difference in POSAS score as assessed by the patient using the Patient Observer Scar Assessment Scale (POSAS) between the treated and untreated half of the scar at 90-days post-treatment compared to baseline. | 90 Days
  The subject will complete the Patient and Observer Scar Assessment Scale (6 questions) prior to treatment and at each follow up visit on both halves of the scar (treated and untreated). Scores will be tabulated and compared for improvement at 90 days after treatment.
3. Patient satisfaction questionnaire at the 90-day follow-up visit. | 90 Days
  Each subject will complete a Patient Satisfaction Questionnaire (PSQ) at the 90 follow-up visit. These results will be tabulated to assess subjects satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Avram, MD, Principal Investigator — MGH Dermatology, Laser and Cosmetic Center
Locations (1):
- MGH Dermatology Laser and Cosmetic Center, Boston, Massachusetts, United States